CLINICAL TRIAL: NCT05206851
Title: Effects of Manual Lymphatic Drainage on Pregnancy Induced Lumbo-Pelvic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Rida Zafar
Record Dates: First submitted 2022-01-21; First posted 2022-01-25 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Low Back Pain
Keywords: low back pain; manual lymphatic drainage; pregnancy
MeSH Terms: conditions — Low Back Pain | interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Lymphatic Drainage and Hot pack (Experimental)
  Interventions: Other: Manual Lymphatic Drainage and Hot Pack
- Hot Pack (Active Comparator)
  Interventions: Other: Hot Pack

INTERVENTIONS:
Other: Manual Lymphatic Drainage and Hot Pack — Application of hot pack for 20 minutes at low back in sitting, and then the participant will perform deep diaphragmatic breathing for 10 minutes, following these steps:
  1. Sitting in comfortable position
  2. One hand is placed over chest and other on abdomen.
  3. Inhale deep through the nose.
  4. Exhale through mouth, completely, counting back from 4 to 1. Application rotary or stationary circle over low back in side lying position, in pregnant females. A session of 20-30 minutes of Manual Lymphatic Drainage will be given biweekly.
  And at the end of Manual Lymphatic Drainage application, deep breathing for 10 minutes will be performed again.
  Arms: Manual Lymphatic Drainage and Hot pack
Other: Hot Pack — Hot pack will be applied at low back, for 20 minutes as home based protocol.
  Arms: Hot Pack

SUMMARY:
This study will be a randomized controlled trial. This study will be conducted in Civil Hospital, Hassan Abdal. A sample size of 32 patients will be taken. Patients will be divided into two groups by lottery method. Group A will be treated with hot pack followed by Manual Lymphatic Drainage while Group B will be given home based plan of hot pack application only. Both groups will receive treatment for 4 weeks,2 sessions per week. The outcome measures Numeric pain rating scale(NPRS), QOL-GRAV and Oswestry Disability Index for back. Data will be analyzed by SPSS 21.

DETAILED DESCRIPTION:
Low back pain is a common complaint among pregnant females. This pain is felt between area of 12th rib and gluteal fold. Pelvic girdle pain(PGP) is proficient among the posterior iliac crest and the gluteal fold, chiefly in the area of the sacroiliac joints and/or in the symphysis pubis. Low back pain is frequent cause for visiting doctor in pregnancy and is related with changed quality of life amongst pregnant females. Health and quality of life of expectant females should be incorporated in the scope of pregnancy routine follow up and precautionary health programs.

Several researchers studied the effect of passive therapeutic techniques to reduce pregnancy induced low back pain. These treatment approaches were compared with active therapeutic techniques (exercise based interventions) or used in combination with active treatment mode to enhance the pain alleviation.

Pregnancy is also associated with lower limb edema due to increase progesterone level that causes blood vessels to relax, making it difficult for blood to return toward heart from lower limb. Most common treatment to reduce edema is Manual Lymphatic Drainage. Manual lymph drainage or Keser I, Esmer M.2019 Manual Lymphatic Drainage is done by a gentle massage on the skin that enhances smooth muscle contraction of the superficial lymphatic vessels and increases the lymphatic flow. Manual Lymphatic Drainage not only reduces edema but also reduce pain along with it. Manual Lymphatic Drainage application is detected by receptors in the skin. It provides the basis of analgesic effect of Manual Lymphatic Drainage. During application of Manual Lymphatic Drainage, numerous adjoining touch receptors are fondled in sequence. Consequently, every receptor directs action potentials at the commencement and termination of the contact, these action potentials prevent the pain.

Drouin JS, Pfalzer L, Shim JM, Kim SJ. 2020 Manual lymph drainage is indicated for reduction of edema of limbs, to reduce pain and fatigue in gravid females. Manual Lymphatic Drainage is also indicated to manage lymphedema succeeding cancer managements and to lessen pain and improve edema instigated by venous ailments, any surgery, and trauma or due to primary lymphedema.

Schingale F-J, Esmer M, Küpeli B, Ünal D. 2021 Manual lymph drainage increase parasympathetic activity and reduce sympathetic activity, increase pain threshold and pain tolerance, improve regeneration and repair of skeletal muscles, increases venous blood recycling, also pain regulation pathway inhibition is Manual Lymphatic Drainage's neural effect.

ELIGIBILITY:
Inclusion Criteria:

* • Expectant female with lumbopelvic pain

  * Posterior pelvic pain
  * Active Straight Leg Raise, Faber, Gaenslen and P4 test positive
  * Pain >3 on NPRS
  * Females in 24- 36 weeks of pregnancy

Exclusion Criteria:

* • Chronic back pain

  * Cellulitis or erysipelas of the treated area
  * Malignant disease of the treated area
  * Disc herniation
  * Lumbar/spinal surgical history
  * Vertebral fracture
  * Acute infection
  * Uncontrolled hypertension
  * High risk pregnancy
  * History of fall or trauma

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 4th week
  NPRS is a segmented version of Visual Analogue Scale (VAS). It consists of number from 0 to 10. Patient selects a number that best reflects his/her pain intensity where 0 is no pain and 10 is maximum pain. For construct validity, NPRS was highly correlated to Visual Analogue Scale (VAS) (0.86-0.95). The test-retest reliability of this scale is recorded to be 0.96. (Hawker et al. 2011)
Quality of Life Questionnaire for Physiological Pregnancy (QOL-GRAV) | 4th week
  The standardized QOL-GRAV questionnaire, focused on assessment of quality of life of pregnant women, was used to gather relevant data and to achieve the goals set. The results of the QOL-GRAV questionnaire are interpreted in such away that the lower the score, the higher the quality of life and the absence of problems associated with speciﬁc changes in pregnancy. The questionnaire assessed 4 domains: physical health, experience, social relationships and the environment .Based on the total score, the quality of life was assessed as excellent, very good, good, or not good.
Oswestry Disability Index for back | 4th week
  The Oswestry Disability Index (also known as the Oswestry Low Back Pain Disability Questionnaire) is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools.

CONTACTS AND LOCATIONS:
Overall Officials: Hadia Nadeem, M.Phil PT, Principal Investigator — Riphah International University
Locations (1):
- Civil Hospital, Hassan Abdal, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No